CLINICAL TRIAL: NCT01032681
Title: A Phase 1, Open-Label, Two-Group, Dose- Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics, Biological and Clinical Activity of EMD 521873 Alone and in Combination With Fixed Low Doses of Cyclophosphamide in Patients With Metastatic or Locally Advanced Solid Tumors or B-Cell Non-Hodgkin Lymphoma
Brief Title: EMD 521873 in Advanced Solid Tumors, MTD Finding
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR62235_001
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2012-10

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Solid tumor; B-Cell Non-Hodgkin Lymphoma; Immunocytokine; interleukin-2; immunotherapy; Metastatic or Locally Advanced Solid Tumors or B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Neoplasm Metastasis | interventions — EMD 521873

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Dose escalation of EMD 521873 monotheraphy 3 doses per cycle
  Interventions: Biological: EMD 521873
- Group 2 (Experimental): Low dose CPA + Dose escalation of EMD 521873 three doses per cycle
  Interventions: Biological: EMD 521873
- Group 3 (Experimental): Dose escalation of EMD 521873 monotheraphy 1 dose per cycle
  Interventions: Biological: EMD 521873

INTERVENTIONS:
Biological: EMD 521873 — Dose escalation steps:
  Group 1: 0,075mg/kg - 0,15mg/kg - 0,225mg/kg - 0,3mg/kg - 0,45mg/kg - 0,6mg/kg - 0,9mg/kg (-1,8mg/kg - 2,1mg/kg - 2,5mg/kg - 3,0mg/kg)
  Disease control and decision of continuation in patient who benefit from the treatment:
  Every second cycle
  Arms: Group 1
Biological: EMD 521873 — Dose escalation steps:
  Group 2: CPA plus 0,6mg/kg - 0,9mg/kg
  Disease control and decision of continuation in patient who benefit from the treatment:
  Every second cycle
  Arms: Group 2
Biological: EMD 521873 — Dose escalation steps:
  Group 3: 0,9mg/kg - 1,2mg/kg - 1,5mg/kg (-1,8mg/kg - 2,1mg/kg - 2,5mg/kg - 3,0mg/kg)
  Disease control and decision of continuation in patient who benefit from the treatment:
  Every second cycle
  Arms: Group 3

SUMMARY:
Primary trial objective in this three arm trial is to assess the safety and tolerability of EMD 521873, and to determine whether the maximum tolerated dose (MTD) is reached with EMD 521873 doses of up to 1.5 mg/kg given alone or in combination with fixed, low-dose cyclophosphamide (CPA) in patients with metastatic or locally advanced solid tumors or B-cell non-Hodgkin lymphoma.

Secondary objectives are to evaluate pharmacokinetic, immunogenicity, overall and best clinical response, changes in tumor marker levels, survival and biological/immune responses to EMD 521873. A total of 78 patients are planned. Patients will remain on the dose throughout the trial. It is intended to administer 3 cycles (21 d each, or until progression or a xxx line therapy becomes necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Male or female, aged ≥ 18 years, inpatient for treatment phase of cycle 1 and 2, outpatient treatment possible for subsequent cycles
3. Histologically or cytologically proven metastatic or locally advanced solid tumors (epithelial or mesenchymal cancers) or B-cell non-Hodgkin lymphoma for which no standard therapy exists or after failure of standard therapy
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at study entry and an estimated life expectancy of at least 3 months
5. Adequate hematological function defined by WBC count ≥ 3 x 109/L with absolute neutrophil count (ANC) ≥ 1.5 x 109/L and lymphocyte count ≥ 0.5 x 109/L; platelet count ≥100 x 109/L; hemoglobin ≥9 g/dL ( If the laboratory values for hemoglobin are outside the required entry level at Screening, a patient may receive a transfusion of RBC. A stable hemoglobin level of ≥9 mg/dL for at least 7 days must be achieved prior to receiving the first dose of study medication.)
6. Adequate hepatic function defined by a total bilirubin level ≤ 1.5 times the upper limit of normal (ULN) and aspartate-aminotransferase (AST) and alanine-aminotransferase (ALT) levels ≤ 2.5 x ULN or, for patients with documented metastatic disease to the liver, AST and ALT levels ≤ 5 x ULN
7. No history of acute or chronic kidney disease and adequate renal function defined by an estimated creatinine clearance above 50 mL/min determined by 24-hour urine sampling or by the Cockcroft-Gault formula
8. Effective contraception for both male and female subjects if the risk of conception exists

Exclusion Criteria:

1. Prior IL-2 therapy within the last 6 months
2. Requirement for concurrent anticancer treatment (chemotherapy, radiotherapy, immune therapy, cytokine therapy except erythropoietin) or for concurrent systemic therapy with steroids or other immunosuppressive agents. Short-term administration of steroids (i.e. for allergic reactions) is allowed.
3. Radiotherapy, chemotherapy, surgery (excluding prior diagnostic biopsy) or any investigational drug in the 30 days before the start of treatment in this study
4. Acquired immune defects such as human immunodeficiency virus (HIV)
5. Systemic autoimmune disease (e.g. lupus erythematodes, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma)
6. Organ transplant recipients
7. History of or active inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis)
8. Chronic viral infections (e.g. hepatitis B virus [HBV], hepatitis C virus [HCV])
9. Uncontrolled hypertension (systolic >180 mmHg, diastolic >100 mmHg)
10. Known hypersensitivity reactions to any of the compounds of the study medication
11. Confirmed or clinically suspected brain metastases
12. Pregnancy (absence to be confirmed by beta-human chorionic gonadotropin [β-HCG] test) or lactation period
13. Clinically significant (i.e. active) cardiovascular disease: Cerebral vascular accident /stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina, congestive heart failure or serious cardiac arrhythmia requiring medication.
14. Pulmonary disease which, in the opinion of the investigator, might impair the patient's respiratory tolerance to moderate pulmonary fluid overload (e.g. interstitial lung disease, severe chronic obstructive pulmonary disease)
15. All conditions which are associated with significant necroses of non tumor-bearing tissues like e.g. esophageal or gastroduodenal ulcers (< 6 months prior to enrolment), organ infarctions (< 6 months prior to enrolment) or active ischemic bowel disease
16. Presence of medically significant third space fluid (pericardial effusion or ascites/ pleural infusion requiring repetitive paracentesis)
17. Known alcohol or drug abuse
18. Participation in another clinical trial within the past 30 days before start of study treatment
19. All other significant diseases which, in the opinion of the investigator, might impair the patient's tolerance of study treatment.
20. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-12; Primary Completion 2011-02 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of EMD 521873 | First administration of any dose of EMD521873 until last administration plus 30 days.
To determine whether the MTD is reached with EMD 521873 doses of up to 1.5 mg/kg given alone or in combination with fixed, low-dose CPA in patients with metastatic or locally advanced solid tumors or B-cell non-Hodgkin lymphoma | Incidence of DLTs occurring during the first cycle of administration of any dose of EMD 521873 given alone on 3 times per cycle (group 1) or with fixed low-dose CPA plus EMD 521873 (group 2) or of EMD 521873 given alone on once per cycle (group 3).

SECONDARY OUTCOMES:
Characterize the PK profile of EMD 521873 alone or in combination with fixed lowdose CPA | Cycle 1-3 of EMD 521873 treatment
Evaluate the immunogenicity of EMD 521873 alone or in combination with CPA measured by the induction of o Specific antibodies against the genetically modified IL-2 o Fc-IL2-specific antibodies o Anti-idiotype antibodies | Every EMD 521873 treatment cycle
Collect evidence of best overall response, changes in serum tumor marker levels and best clinical response after treatment with EMD 521873 alone or in combination with CPA | Every second EMD 521873 treatment cycle
Evaluate survival | Until 1 year after the last patient received his last dose of EMD 521873
Evaluate biological responses to EMD 521873 alone or in combination with CPA as measured by o Absolute cell numbers and ratios of lymphocyte subsets in defined combinations o Change in serum level of sIL2R and neopterin | Cycle 1-3 of EMD 521873 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Peter Marschner, MD, Study Director — Merck KGaA, Darmstadt, Germany
Locations (5):
- Germany (2):
  - Universitäts-Klinikum Mainz III.Medizinische Klinik, Mainz
  - Medizinische Klinik Universitätsklinikum Mannheim Medizinische Fakultät Mannheim, Mannheim
- Switzerland (3):
  - Istituto Oncologico della Svizzera Italiana Ospedale Regionale Bellinzona e Valli (IOSI), Bellinzona
  - University of Lausanne Hospitals (CHUV) and Hospitals of Riveria-Chablais, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen